CLINICAL TRIAL: NCT01721603
Title: A Phase 2 Prospective Trial of Dabrafenib and Trametinib With Stereotactic Radiosurgery in BRAF Mutant Melanoma Brain Metastases
Brief Title: Dabrafenib and Trametinib With Radiosurgery in Melanoma Brain Mets
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of California, San Francisco (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Alain Algazi, Assistant Clinical Professor, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12857
Record Dates: First submitted 2012-11-01; First posted 2012-11-06 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: BRAFV600E Melanoma Patients
Keywords: BRAFV600E melanoma patients; melanoma; stereotactic radiosurgery; BRAFV600E melanoma brain metastases; dabrafenib; SRS
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; Radiosurgery; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dabrafenib + Trametinib + gamma knife radiosurgery (Experimental)
  Interventions: Drug: Dabrafenib; Procedure: Gamma Knife Radiosurgery; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — 150 mg capsule by mouth twice daily
  Other Names: GSK2118436
Procedure: Gamma Knife Radiosurgery — This will be delivered using Gamma Knife technology. Patients will be fitted with a stereotactic head-frame for stereotactic localization of brain metastases.
  Other Names: SRS; Stereotactic Radiosurgery
Drug: Trametinib — 2 mg by mouth once daily from beginning at Cycle 3 Day 1, until progression of disease, withdrawal of consent, or the development of intolerable treatment associated toxicity.
  Other Names: GSK1120212

SUMMARY:
The purpose of this study is to test the safety and find out what effects, good and/or bad, dabrafenib (a BRAF inhibitor) alone or dabrafenib when given in combination with gamma knife radiosurgery has on participants with a certain type of skin cancer (BRAFV600E melanoma) and brain metastases (tumors that have spread to the brain).

DETAILED DESCRIPTION:
This is a single arm Phase II clinical trial. All patients will receive continuous dosing of dabrafenib at 150 mg PO bid and trametinib beginning at Cycle 3 Day 1, at a starting dose of 2 mg PO once daily until progression of disease, withdrawal of consent, or the development of intolerable treatment associated toxicity. An MRI will be performed after 28 days of treatment with dabrafenib. Patients who have unequivocal disease progression in the brain at that time will be deemed to have disease progression at 4 weeks. Patients with a complete response of all lesions in the brain will continue to receive dabrafenib and trametinib on study but they will not undergo SRS. For patients with stable disease or partial tumor responses in the brain, Gamma Knife radiosurgery will be performed on treatment cycle 2, day 1 (+/- 3 days, 28 day cycle) using a stereotactic head frame and MRI imaging in accordance with FDA-approved procedures.

Melanoma brain metastases

Cutaneous melanoma is the most aggressive form of all skin cancers. Worldwide, it is currently expected that approximately 132,000 people will be diagnosed with melanoma each year and some 37,000 people are expected to die of the disease annually. Brain metastases are a major source of morbidity and mortality in patients with metastatic melanoma and approximately 3 out of 4 develop brain metastases at some point in their disease course. The prognosis of metastatic melanoma with CNS involvement is dismal1, and, until recently, no medical therapy demonstrated clear evidence of activity against melanoma in the brain. For patients with fewer than 4 brain lesions and no brain lesion greater than 3 cm in diameter, stereotactic radiosurgery (SRS) is the standard-of-care. By delivering highly focal irradiation to melanoma brain metastases, SRS confers local control rates exceeding 80% for lesions under 2 cm in diameter. However, SRS does not treat micrometastatic disease in the brain, and new brain metastases develop in approximately half of patients treated.

Furthermore, local control rates are lower for lesions larger than 2 cm in diameter. As a result, the median overall survival for melanoma patient treated with SRS is only 7 months.

BRAF mutant melanoma

The RAS/RAF/MEK/ERK pathway is a critical proliferation pathway in many human cancers. This pathway can be constitutively activated by alterations in specific proteins, including BRAF, which phosphorylates MEK1 and MEK2 on two regulatory serine residues. Approximately 90% of all identified BRAF mutations that occur in human result in a V600 E/D/Kamino acid substitution. This mutation appears to mimic regulatory phophorylation and increases BRAF activity approximately 10-fold compared to wild type. BRAF mutations have been identified at a high frequency in specific cancers, including approximately 40-60% of melanoma. The frequency of this activating mutation and the pathway addiction to which it leads makes mutated BRAF an extremely attractive target.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed BRAFV600E melanoma
2. Up to 4 untreated brain metastases (at least 1 > 0.5 cm) with no metastasis larger than 3 cm as assessed by a gadolinium-enhanced MRI of the brain. Detection of additional lesions at time of Gamma Knife radiosurgery MRI scan will not be considered exclusionary if the detection of these lesions are thought to be due solely to difference in imaging techniques (i. e. higher sensitivity, double gadolinium contrast MRI utilized at the time of Gamma Knife radiosurgery compared with conventional MRI imaging).
3. ECOG PS 0-2
4. 14 days elapsed from last treatment with surgery.
5. At least 28 days or five half-lives (whichever is longer) have elapsed from last dose of any approved or investigational therapy for metastatic melanoma.
6. Appropriate birth control for men and women with childbearing potential
7. Corticosteroid dose stable for at least 14 days
8. Adequate end-organ function:

   * ANC ≥ 1.5x109/L
   * Hemoglobin ≥ 9 g/dL
   * Platelets ≥100 x109/L
   * Total bilirubin ≤ 1.5x ULN
   * AST and ALT ≤ 2.5x ULN
   * Creatinine ≤ 1.5 mg/dL
   * PT/PTT ≤ 1.5x ULN
   * LVEF ≥ 50%
9. Age ≥ 18 years
10. Recipients of prior radiation therapy to the brain including stereotactic radiosurgery or whole brain irradiation may be included if there are 1-4 untreated or progressing brain lesions. At his discretion, the Study Chair may review any enrollment decision regarding which subjects will be enrolled prior to the initiation of treatment on trial.

Exclusion Criteria:

1. Neurological symptoms from melanoma brain metastases
2. Patients may not have received prior therapy with dabrafenib, vemurafenib, or other potent, highly effective BRAF inhibitors. Prior therapy with sorafenib is permitted.
3. Any indication for urgent or emergent neurosurgery. Patient may enroll after neurosurgery at least 14 days after neurosurgery as long as they meet all other study qualifications.
4. Pregnant or lactating women. The effects of dabrafenib on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use a highly effective method of contraception including: hormonal contraceptives (oral contraceptives, Nuvaring, Depo Provera) an intrauterine device, true abstinence or two barrier methods of birth control including condoms with cervical cap or diaphragm. Baseline pregnancy testing is required for all women of child-bearing potential. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol who are sexually active with women of child bearing potential must also agree to use adequate contraception prior to and during the study as outlined above, and for, and four months after completion of study drug administration.
5. History of known cardiac arrhythmias or acute coronary syndromes within the past 24 weeks.
6. History of a second malignancy with evidence of active disease within the past 3 years except non-melanoma skin cancer, indolent prostate cancer, and stable CLL without lymphadenopathy
7. Complete resection of a single brain metastasis or of all known brain metastases. Patients who have undergone subtotal resection are eligible providing residual disease is < 2.0 cm in maximum diameter.
8. Patients with metastases within 2 mm of the optic nerve or optic chiasm so that some portion of the optic nerve or chiasm would receive > 9 Gy from radiosurgery.
9. Patients with metastases in the brainstem.
10. Contraindication to MRI (such as cardiac pacemaker).
11. The following medications or non-drug therapies are prohibited:

    * Other anti-cancer therapy while on treatment in this study.
    * Use of other investigational drugs within 28 days preceding the first dose of dabrafenib.
    * Antiretroviral drugs. Subjects with known HIV are ineligible for study participation.
    * Herbal remedies (i.e., St. John's wort).
    * Drugs that are strong inhibitors or inducers of CYP3A or CYP2C8, p-glycoprotein (Pgp) or Bcrp transporter because they may alter dabrafenib concentrations. The list may be modified based on emerging data. These include but are not limited to those listed in Appendix 2; consider therapeutic substitutions for these medications.
12. Unresolved toxicity of National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0. Grade 2 or higher from previous anti-cancer therapy, except alopecia.
13. Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption of drugs. If clarification is needed as to whether a condition will significantly affect absorption of drugs, contact the Study Chair for permission to enroll the subject. Study Chair has final decision regarding which subjects will be enrolled.
14. A history of known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection. Subjects with laboratory evidence of HBV clearance may be enrolled with permission of the GSK medical monitor.
15. A history of known glucose-6-phosphate dehydrogenase (G6PD) deficiency.
16. Corrected QT (QTc) interval ≥480 msecs; history of acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting within the past 24 weeks; Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system; abnormal cardiac valve morphology documented by echocardiogram (subjects with minimal abnormalities including mild regurgitation/stenosis can be entered on study with approval from the GSK medical monitor); or history of known cardiac arrhythmias.
17. Treatment refractory hypertension defined as a blood pressure of systolic> 140 mmHg and/or diastolic > 90 mm Hg which cannot be controlled by anti-hypertensive therapy.
18. History of RVO or CSR, or predisposing factors to RVO or CSR(e.g. uncontrolled glaucoma or ocular hypertension, uncontrolled systemic disease such as diabetes mellitus, hypertension, or history of hyperviscosity or hypercoagulability syndromes)
19. Visible retinal pathology as assessed by ophthalmic exam that is considered a risk factor for RVO or CSR such as:

    * Evidence of new optic disc cupping
    * Evidence of new visual field defects
    * Intraocular pressure > 21 mm Hg as measured by tonography
20. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol; or unwillingness or inability to follow the procedures required in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alain Algazi, MD, Study Chair — University of California, San Francisco
Locations (1):
- University of San Francisco, California, San Francisco, California, United States

REFERENCES:
- [Derived] Patel KR, Chowdhary M, Switchenko JM, Kudchadkar R, Lawson DH, Cassidy RJ, Prabhu RS, Khan MK. BRAF inhibitor and stereotactic radiosurgery is associated with an increased risk of radiation necrosis. Melanoma Res. 2016 Aug;26(4):387-94. doi: 10.1097/CMR.0000000000000268. PMID 27223498

RESULTS

PARTICIPANT FLOW:
Groups:
- Dabrafenib + Trametinib + Gamma Knife Radiosurgery: 1 cycle = 28 days
  * Dabrafenib: 150mg capsule by mouth (PO), twice daily, continuous
  * Trametinib: 2 mg PO, once daily from beginning of cycle 3 Day 1,until progression of disease, withdrawal of consent, or the development of intolerable treatment associated toxicity.
  For patients with stable disease or partial tumor responses in the brain, Gamma Knife radiosurgery will be performed on treatment cycle 2, day 1 (+/- 3 days) using a stereotactic head frame and MRI imaging in accordance with FDA-approved procedures.
Period: Overall Study
Arm/Group | Dabrafenib + Trametinib + Gamma Knife Radiosurgery
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Dabrafenib Given in Combination With Gamma Knife Radiosurgery: All patients will receive continuous, oral dosing of dabrafenib at a starting dose of 150 mg twice daily until progression of disease, withdrawal of consent, or the development of intolerable treatment associated toxicity
  Dabrafenib: 150mg capsule by mouth twice daily
  Gamma Knife Radiosurgery: This will be delivered using Gamma Knife technology. Patients will be fitted with a stereotactic head-frame for stereotactic localization of brain metastases.
Arm/Group | Dabrafenib Given in Combination With Gamma Knife Radiosurgery
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Patients Reaching 6 Month Distant Brain Metastasis-free Survival (DBMFS)
Description: Determine whether dabrafenib combined with stereotactic radiosurgery (SRS) and trametinib improves the 6 month DBMFS rate of BRAFV600E melanoma patients for whom the standard of care is stereotactic radiosurgery (≤4 brain lesions and no lesion > 3 cm) in comparison with similar historical controls treated with radiosurgery alone.
Time Frame: Up to 6 months after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib + Trametinib + Gamma Knife Radiosurgery
Number analyzed (Participants) | 2
Participants | 1

2. Secondary Outcome: Patients Displaying 6-month Local Control Rate
Description: Determine whether dabrafenib combined with SRS and trametinib improves the 6-month local control rate of BRAFV600E melanoma brain metastases compared with historical controls treated with SRS.
Time Frame: From surgery up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib + Trametinib + Gamma Knife Radiosurgery
Number analyzed (Participants) | 2
Participants | 1

3. Secondary Outcome: Best Overall Response Rate (by RECIST v1.1 )
Description: Determine the best overall response rate (by RECIST v1.1 ).
Time Frame: From surgery up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib + Trametinib + Gamma Knife Radiosurgery
Number analyzed (Participants) | 2
Participants | 1

4. Secondary Outcome: Median Duration of Freedom From New Brain Metastases( by RECIST v1.1 )
Description: Determine median duration of freedom from new brain metastases of BRAFV600E melanoma brain metastases patients treated with SRS, trametinib and dabrafenib. RECIST v1.1 will be used as the primary determinant of disease progression.
Time Frame: From surgery up to 12 months
Population: Study was terminated due to low accrual. Secondary outcome measure was not accessed.
Arm/Group | Dabrafenib + Trametinib + Gamma Knife Radiosurgery
Number analyzed (Participants) | 0

5. Secondary Outcome: Median Time to Progression
Description: Determine the median time to progression in the brain of BRAFV600E melanoma brain metastases patients treated with SRS, trametinib and dabrafenib. RECIST v1.1 will be used as the primary determinant of disease progression. Disease response will be assessed at scheduled visits by MRI of the brain and clinical exam every two months thereafter. The proportion of patients that progression free at 6 months will be calculated.
Time Frame: From surgery up to 12 months
Population: Study was terminated due to low accrual. Secondary outcome measure was not accessed.
Arm/Group | Dabrafenib + Trametinib + Gamma Knife Radiosurgery
Number analyzed (Participants) | 0

6. Secondary Outcome: Systemic Overall Response Rate
Description: Determine the systemic best overall response rate of BRAFV600E melanoma brain metastasis patients treated with SRS, trametinib and dabrafenib.
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
  The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that recurrent disease is objectively documented.
Time Frame: From surgery up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib + Trametinib + Gamma Knife Radiosurgery
Number analyzed (Participants) | 2
Participants | 1

7. Secondary Outcome: Median Progression-free Survival
Description: Determine the median progression-free survival of BRAFV600E melanoma brain metastasis patients treated with SRS, trametinib and dabrafenib.
Time Frame: From surgery up to 12 months
Population: Study was terminated due to low accrual. Secondary outcome measure was not accessed.
Arm/Group | Dabrafenib + Trametinib + Gamma Knife Radiosurgery
Number analyzed (Participants) | 0

8. Secondary Outcome: Median Overall Survival
Description: Determine the median overall survival of BRAFV600E melanoma brain metastasis patients treated with SRS, trametinib and dabrafenib.
Time Frame: From surgery up to 12 months
Population: Study was terminated due to low accrual. Secondary outcome measure was not accessed.
Arm/Group | Dabrafenib + Trametinib + Gamma Knife Radiosurgery
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Dabrafenib With Gamma Knife Radiosurgery: Dabrafenib: 150mg capsule by mouth twice daily until progression of disease, withdrawal of consent, or the development of intolerable treatment associated toxicity
  Gamma Knife Radiosurgery: This will be delivered using Gamma Knife technology. Patients will be fitted with a stereotactic head-frame for stereotactic localization of brain metastases.
Arm/Group | Dabrafenib With Gamma Knife Radiosurgery
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabrafenib With Gamma Knife Radiosurgery (N=2)
Fatigue (General disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Flushing (Vascular disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Headache (Nervous system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Anxiety (Psychiatric disorders) | 1
Nipple hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Fever (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Malaise (General disorders) | 1
Rhinorrhea (Skin and subcutaneous tissue disorders) | 1
External ear canal hyperkeratosis (Ear and labyrinth disorders) | 1
Foot pain (Musculoskeletal and connective tissue disorders) | 1
Hand foot reaction (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes